CLINICAL TRIAL: NCT00444249
Title: Influence of Blue Light Filtering Intra Ocular Lenses on Daytime Levels of Melatonin in Patients With Non-Exudative Age-Related Macular Degeneration
Brief Title: Influence of Blue Light Filtering Intraocular Lenses on Daytime Levels of Melatonin
Acronym: BluMel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because only a few patients follow the inclusion and exclusion criteria.
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Prof. Dr. Susanne Binder, Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LBI-06-172-1006
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Macular Degeneration
Keywords: age-related macular degeneration; melatonin; blue-light filter
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): White Alcon IOL
  Interventions: Procedure: White Alcon IOL
- 2 (Active Comparator): Yellow Alcon IOL
  Interventions: Procedure: Yellow Alcon IOL
- 3 (Active Comparator): White Hoya IOL
  Interventions: Procedure: White Hoya IOL
- 4 (Active Comparator): Yellow Hoya IOL
  Interventions: Procedure: Yellow Hoya IOL

INTERVENTIONS:
Procedure: White Alcon IOL — Implantation of white Alcon IOL
  Arms: 1
Procedure: Yellow Alcon IOL — Implantation of yellow Alcon IOL
  Arms: 2
Procedure: White Hoya IOL — Implantation of white Hoya IOL
  Arms: 3
Procedure: Yellow Hoya IOL — Implantation of yellow Hoya IOL
  Arms: 4

SUMMARY:
The "blue light hazard" has been reported to cause retinal damage (oxidative stress), particularly to the central fovea due to its energetic, shorter wavelength visible photons, which is why blue-light filtering intraocular lenses have been developed for cataract surgery. The hormone melatonin has been reported to possess an efficient antioxidant capacity. Light information from the eye reaches the suprachiasmatic nuclei and inhibits melatonin secretion. Since melatonin is suppressed by light, we have a day-night rhythmicity, with increased levels at night. Melatonin suppression is wavelength-dependent with a peak sensitivity in the 446-477 nm (blue light) portion of the visible spectrum. The crystalline lens blocks most UV between 300 and 400 nm. The density of the lens increases with aging causing an alteration in the spectral absorption. The greatest increase in absorption occurs at the short wavelength end of the spectrum (around 400-470 nm). Age-related pupillary miosis and crystalline lens yellowing limit the blue light reaching the retina. This reduces the older adults' effective retinal light exposure to one tenth that of younger people. It has been shown that insomnia and depression decrease after cataract surgery and patients returned to youthful levels of melatonin. Since melatonin acts as an antioxidant, and more blue light filtering intra ocular lenses are implanted and thought to reduce photochemical damage in the macula, it would be interesting to show the positive influence of those blue light filtering intraocular lenses on daytime levels of melatonin in age-related macular degeneration patients.

DETAILED DESCRIPTION:
Patients with non-exudative age-related macular degeneration, which are planned for cataract surgery, will be randomized into one of four groups. Group I and II are blue light filtering intraocular lenses and group III and IV are white lenses. Group I and III are lenses form Alcon, group II and IV are lenses form Hoya. The following examinations will be performed before, 1 month, 6 months, 1 year and 2 years after surgery: vein puncture for melatonin analysis, visual acuity, complete slit lamp analysis including intraocular pressure, pupil size measurement, and questionnaire about sleeping time and sleeping quality. At the follow-up visits the following examinations will also be performed: autofluorescein imaging, infrared imaging, and optical coherence tomography imaging. Vein puncture will be performed between 8 and 10 a.m. and has to be performed at the same time for the same patient. Pupils are not allowed to be dilated by the time of vein puncture and pupil size measurement.

ELIGIBILITY:
Inclusion Criteria:

Patients are included if they meet all of the following inclusion criteria:

* Cataract on one or both eyes
* Study eye with non-exudative AMD AREDS I - III
* Men or women aged between 60 - 99 years
* Patient planned for cataract surgery and in need of an intraocular lens

Exclusion Criteria:

Patients are excluded if they meet one or more of the following exclusion criteria:

* Study eye with exudative AMD
* Study eye with concomitant retinal or choroidal disorder other than AMD
* Study eye with significant keratopathies
* Fundus not visible
* Intake of medication known to affect melatonin secretion (within the last 12 hours): ß-blockers, calcium channel blockers, a-blockers, non-steroidal anti-inflammatory drugs, benzodiazepines, antidepressants, hypnotic drugs, antipsychotics, barbiturates, antiepileptic drugs, and melatonin
* Alcohol or caffeine consumption 6 hours before vein puncture
* Patients who are unwilling to adhere to visit examination schedules

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Melatonin daytime levels in serum | 1, 6, 12, and 36 months postoperative

SECONDARY OUTCOMES:
Number of drusen, retinal thickness, pupil size, sleeping time | 1, 6, 12, and 36 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Katharina E. Schmid-Kubista, MD, Principal Investigator — LBI
Locations (1):
- Rudolf Foundation Clinic, Department of Ophthalmology, Vienna, Vienna, Austria